CLINICAL TRIAL: NCT02135575
Title: Effects of Exercise Training on Cardiovascular Health in Middle-aged Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Glostrup University Hospital, Copenhagen (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Ylva Hellsten, Professor, University of Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CWS-WP2CV
Record Dates: First submitted 2014-04-01; First posted 2014-05-12 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Menopause; Cardiac Function Impaired; Cardiovascular Diseases; Blood Platelet Disorders; Metabolic Diseases
Keywords: premenopausal; postmenopausal; cardiovascular; exercise training; vascular function; cardiac function; cardiac morphology; health
MeSH Terms: conditions — Cardiovascular Diseases; Blood Platelet Disorders; Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Premenopausal women (Experimental): The Premenopausal women are randomized to exercise by spinning (cycle)
  Interventions: Behavioral: Spinning
- Postmenopausal women (Experimental): The Postmenopausal women are randomized to exercise by spinning (cycle)
  Interventions: Behavioral: Spinning

INTERVENTIONS:
Behavioral: Spinning — After the baseline studies the pre and postmenopausal women will be randomized to spinning training groups and the intervention will last for 3 months. The spinning group will spin three times per week under guidance of a trained instructor. The training is heart rate monitored.

SUMMARY:
The hypothesis of the present study is that physical training can oppose detrimental changes in cardiovascular and metabolic health associated with estrogen loss after menopause.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal (45-53 years) OR postmenopausal 50-57 years
* BMI> 18.5 and <30
* Sedentary (no regular physical activity the last 2 years)
* Plasma measurements
* Premenopausal: estradiol> 0.20 nmol/l, Follicle stimulating hormone < 22 IU/l and progesterone >2.5 nmol/l
* Postmenopausal: estradiol < 0.20 nmol/l, Follicle stimulating hormone > 22 IU/l and progesterone 0.3-2.5 nmol/l

Exclusion Criteria:

* Smoking
* Excessive alcohol intake
* Regular medication including hormone replacement treatment
* Chronic disease

Ages: 45 Years to 57 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2014-05; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Leg vascular function | Baseline comparison and changes from baseline to 3 months
  Measurements of leg blood flow by ultrasound doppler during exercise and during femoral arterial infusion of vasodilators
Cardiac structure and function | Baseline comparison and changes from baseline to 3 months
  Magnetic resonance imaging and transthoracic echocardiography
Platelet function | Baseline comparison and changes from baseline to 3 months
  Platelet aggregation assay of whole blood and platelet rich plasma

SECONDARY OUTCOMES:
Expression of proteins in muscle samples | Baseline comparison and changes from baseline to 3 months
  Western Blot analysis of proteins of relevance for vascular function and metabolism
Maximal aerobic effect | Baseline comparison and changes from baseline to 3 months
  Maximal oxygen uptake during an incremental cycle ergometry test with gas analysis
Genomic profile in blood samples | Baseline comparison and changes from baseline to 3 months
  Genomic analysis of parameters for vascular and metabolic health
Insulin sensitivity and glycaemic control | Baseline comparison and changes from baseline to 3 months
  Fasting plasma glucose analysis and oral glucose tolerance test
Arterial blood pressure | Baseline comparison and changes from baseline to 3 months
Gene expression of proteins in muscle samples | Baseline comparison and changes from baseline to 3 months
  Gene analysis of relevance for vascular and metabolic function
Health related parameters in blood | Baseline comparison and changes from baseline to 3 months
  Plasma lipid status and other variables related to vascular health

OTHER OUTCOMES:
Anthropometry | Baseline comparison and changes from baseline to 3 months
  Dual x-ray absorptiometry, height, weight, waist and hip circumference
Activity measure | Baseline comparison and changes from baseline to 3 months
  Activity measure for one week by accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: Erik Richter, MD PhD, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Egelund J, Jorgensen PG, Mandrup CM, Fritz-Hansen T, Stallknecht B, Bangsbo J, Nyberg M, Hellsten Y. Cardiac Adaptations to High-Intensity Aerobic Training in Premenopausal and Recent Postmenopausal Women: The Copenhagen Women Study. J Am Heart Assoc. 2017 Aug 18;6(8):e005469. doi: 10.1161/JAHA.117.005469. PMID 28862950